CLINICAL TRIAL: NCT02292212
Title: Clinical Study of Asahi ViE Dialyzer in Canada (AVID)
Brief Title: Clinical Study of Asahi ViE Dialyzer in Canada
Acronym: AVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asahi Kasei Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVID
Record Dates: First submitted 2014-10-28; First posted 2014-11-17 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): The dialyzer will be changed from conventional one to ViE-21 for 36 sessions for all the enrolled subjects.
  Interventions: Device: ViE-21

INTERVENTIONS:
Device: ViE-21 — The subjects will be undergone three times KUF measurement sessions and three times blood sampling sessions during study period.

SUMMARY:
The purpose of the study is to obtain performance data on the Asahi ViE-21 dialyzer (ViE-21) .

DETAILED DESCRIPTION:
The objective of the study is to evaluate specific parameters related to ViE-21 performance including (A) Performance evaluated by uremic solute removal rates of urea, creatinine, albumin and B2-MG, (B) Determination of KUF, (C) Biocompatibility evaluated by WBC, platelet and C3a measurements, (D) Type and number of adverse events, (E) Type and number of device malfunctions.

Prospective, open-label, non-randomized, single-armed, controlled study. Each patient shall have data collected for six dialysis sessions each on a control dialyzer prior to and after 36 sessions with the ViE-21. These data shall be the basis of comparison for the ViE-21 performance.

These data will be utilized in support of a US Regulatory Submission.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years and ≤ 80 years of age
2. Stable on maintenance hemodialysis for at least 12 weeks
3. Patients expected to remain on hemodialysis for at least 24 weeks
4. Patients on hemodialysis for more than 3 hours per treatment and on a 3 times per week schedule
5. Patients whose vascular access is obtained via arteriovenous fistula or graft, is well maintained and is capable of obtaining blood flow rate ≥ 350 mL/min during the study period
6. Patients using high-flux dialyzers (KUF ≥ 40 mL/hr/mmHg) with surface area ≥ 1.5 square meters and ≤ 2.2 square meters
7. Patients capable of understanding the informed consent form
8. Written consent and willingness to participate in the study

Exclusion Criteria:

1. Medical conditions requiring regular blood transfusion
2. Patients with a history of more than one week hospitalization related to infection, inflammation or surgery within the past 12 weeks
3. Patients having participated in another clinical investigation within the past 12 weeks, currently participating or having a plan of participating in any other clinical investigation (patients in an observational study without any interventions or in post-market surveillance do not need to be excluded)
4. Patients who have difficulty in maintaining vascular access function within the past 12 weeks
5. Patients who are known to be hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) positive
6. Female patients who are pregnant, breast feeding or planning a pregnancy within the study period
7. Patients having received blood purification therapy other than conventional dialysis within the past 12 weeks
8. Patients who cannot tolerate Heparin
9. Any serious medical, social or psychological condition that in the opinion of the investigator would disqualify a patient from participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2015-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedeh Kiaii, MD, Principal Investigator — St. Pauls Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiaii M, Aritomi M, Nagase M, Farah M, Jung B. Clinical evaluation of performance, biocompatibility, and safety of vitamin E-bonded polysulfone membrane hemodialyzer compared to non-vitamin E-bonded hemodialyzer. J Artif Organs. 2019 Dec;22(4):307-315. doi: 10.1007/s10047-019-01110-w. Epub 2019 Jun 26. PMID 31254226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients on hemodialysis at one clinical site in Canada were enrolled to this study. The first patient was enrolled on November 24, 2014 and the last patient on July 13, 2015.
Groups:
- Single Arm: Total 16 weeks, divided to 3 periods, Pre-ViE phase (2W by control device), ViE phase (12W by target device, ViE-21) and Post-ViE phase (2W by control device).
Period: Pre-ViE Phase
Arm/Group | Single Arm
Started | 17
Completed | 17
Not Completed | 0
Period: ViE Phase
Arm/Group | Single Arm
Started | 17
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Period: Post-ViE Phase
Arm/Group | Single Arm
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Total 16 weeks, divided to 3 phases, Pre-ViE phase (2W by control device), ViE phase (12W by target device, ViE-21) and Post-ViE phase (2W by control device).
Arm/Group | Single Arm
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7
  Black or African American | 0
  Asian | 2
  Hispanic | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Asian Filipino | 4
  Asian Indian | 2
  Asian Sri Lankan | 1
  Native Canadian | 1

OUTCOME MEASURES:

1. Primary Outcome: Removal Rate of Urea
Description: In order to calculate removal rate for urea by a dialysis session, blood samples were collected at pre and post dialysis. The removal rate was obtained by calculation using the following equation with Pre-dialysis concentration (Cpre) and Post-dialysis concentration (Cpost) of urea.
  Removal rate (%) = [(Cpre - Cpost) / (Cpre)] * 100. The removal rates were obtained at one session of the first week with control dialyzer (Pre-ViE phase) and then at each one session of weeks 7 and 13 with ViE-21 (ViE phase), respectively.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of urea removal
Groups:
- Pre-ViE Phase: The first week of dialysis with control dialyzer
- ViE Phase (1): Seventh week of dialysis with ViE-21
- ViE Phase (2): 13th week of dialysis with ViE-21
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of urea removal | 76.1 (5.4) | 74.4 (8.8) | 73.5 (4.5)

2. Primary Outcome: Removal Rate of Creatinine
Description: In order to calculate removal rate for creatinine by a dialysis session, blood samples were collected at pre and post dialysis. The removal rate was obtained by calculation using the following equation.
  Removal rate (%) = [(Cpre - Cpost) / (Cpre)] * 100. The removal rates were obtained at one session of the first week with control dialyzer (Pre-ViE phase) and then at each one session of weeks 7 and 13 with ViE-21 (ViE phase), respectively.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of creatinine removal
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of creatinine removal | 70.7 (4.6) | 70.0 (8.4) | 69.0 (5.4)

3. Primary Outcome: Removal Rate of Albumin
Description: In order to calculate removal rate for albumin by a dialysis session, blood samples were collected at pre and post dialysis. The removal rate was obtained by calculation using the following equation with hematocrit (HCT) at pre (HCTpre) and post (HCTpost).
  Removal rate (%) = {1-[HCTpre*(1-HCTpost/100) * Cpost] / [HCTpost * (1-HCTpre/100) * Cpre]} * 100.
  The removal rates were obtained at one session of the first week with control dialyzer (Pre-ViE phase) and then at each one session of weeks 7 and 13 with ViE-21 (ViE phase), respectively. The negative removal rate means the increase of serum concentration of albumin from pre to post dialysis session.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of albumin removal
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of albumin removal | 2.4 (6.4) | -2.4 (3.9) | -1.0 (4.4)

4. Primary Outcome: Removal Rate of Beta-2-microglobulin (B2-MG)
Description: In order to calculate removal rate for B2-MG by a dialysis session, blood samples were collected at pre and post dialysis. The removal rate was obtained by calculation using the following equation.
  Removal rate (%) = {1-[HCTpre*(1-HCTpost/100) * Cpost] / [HCTpost * (1-HCTpre/100) * Cpre]} * 100.
  The removal rates were obtained at one session of the first week with control dialyzer (Pre-ViE phase) and then at each one session of weeks 7 and 13 with ViE-21 (ViE phase), respectively.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of B2MG removal
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of B2MG removal | 65.5 (6.6) | 65.8 (8.8) | 65.9 (6.5)

5. Primary Outcome: Ultrafiltration Coefficient (KUF)
Description: The KUF is important for regulating the rate and amount of fluid flow across the dialyzer membrane. It is calculated by dividing ultrafiltration rate with the transmembrane pressure (TMP). More specifically, transmembrane pressures were recorded at 10, 20, 30, 40 and 50 minutes after the initiation of the dialysis session with adjustment of the ultrafiltration rate at 0, 600, 1000, 1400 and 1800 mL/hr respectively. These determinations were made during the 2nd or 3rd treatment session during the 1st or 2nd week for control dialyzer (Pre-ViE phase), and for ViE-21 during week 3-8 and week 9-14 (ViE phase).
Time Frame: Week 1 or 2 (Pre-ViE phase), 3-8 and 9-14 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: mL/(hr*mmHg)
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
mL/(hr*mmHg) | 61.2 (13.6) | 67.8 (8.6) | 68.6 (9.3)

6. Primary Outcome: White Blood Cell (WBC)
Description: Blood samples were obtained during the first week of dialysis with control dialyzer and then during weeks 7 and 13 with ViE-21. WBC count was measured pre dialysis, at 15 minutes and post dialysis. The values were corrected with HCT and then leveled by defining the pre-dialysis value as 100%.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of WBC level
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of WBC level
  15 min | 82.3 (13.1) | 86.5 (9.8) | 92.7 (8.0)
  Post dialysis | 95.1 (12.1) | 94.1 (12.4) | 97.1 (12.3)

7. Primary Outcome: Platelet
Description: Blood samples were obtained during the first week of dialysis with control dialyzer and then during weeks 7 and 13 with ViE-21. Platelet count was measured pre dialysis, at 15 minutes and post dialysis. The values were corrected with HCT and then leveled by defining the pre-dialysis value as 100%.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of platelet level
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of platelet level
  15 min | 94.6 (8.5) | 98.4 (4.6) | 98.2 (3.7)
  Post dialysis | 93.9 (8.4) | 99.0 (7.4) | 99.8 (7.5)

8. Primary Outcome: Activated Complement Factor III (C3a )
Description: Blood samples were obtained during the first week of dialysis with control dialyzer and then during weeks 7 and 13 with ViE-21. C3a was measured pre dialysis, at 15 minutes and post dialysis. The values were corrected with HCT and then leveled by defining the pre-dialysis value as 100%.
Time Frame: Week 1 (Pre-ViE phase), 7, 13 (ViE phase)
Population: The Intent To Treat (ITT) was based on 14 patients that received at least 30 treatments with ViE-21.
Measure: Mean (Standard Deviation); unit: percentage of C3a level
Arm/Group | Pre-ViE Phase | ViE Phase (1) | ViE Phase (2)
Number analyzed (Participants) | 14 | 14 | 14
percentage of C3a level
  15 min | 224.1 (112.2) | 236.2 (115.2) | 198.1 (99.2)
  Post dialysis | 97.3 (29.5) | 103.1 (29.2) | 90.2 (33.7)

9. Secondary Outcome: Device Malfunctions
Time Frame: Week 1 to 2 (Pre-ViE phase), 3 to 14 (ViE phase), and 15 to 16 (Post-ViE phase)
Population: The safety analysis population (SAA) that is comprised of all patients that received at least one session with the ViE-21
Measure: Number; unit: malfunctions
Groups:
- Pre-ViE Phase: Two weeks (six sessions) on the control dialyzer
- ViE Phase: 12 weeks (36 sessions) on the ViE-21
- Post ViE Phase: Two weeks (six sessions) on the same model control dialyzer used during the pre-ViE phase
Arm/Group | Pre-ViE Phase | ViE Phase | Post ViE Phase
Number analyzed (Participants) | 17 | 17 | 14
malfunctions | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Two weeks for Pre-ViE phase, 12 weeks for ViE phase and 2 weeks for Post-ViE phase
Groups:
- Pre-ViE Phase: Two weeks (six sessions) on control dialyzer
- ViE Phase: 12 weeks (36 sessions) on ViE-21
- Post-ViE Phase: Two weeks (six sessions) on the same model control dialyzer used during the pre-ViE phase
Arm/Group | Pre-ViE Phase | ViE Phase | Post-ViE Phase
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 1/14
Other Adverse Events (participants affected / at risk) | 16/17 | 17/17 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-ViE Phase (N=17) | ViE Phase (N=17) | Post-ViE Phase (N=14)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-ViE Phase (N=17) | ViE Phase (N=17) | Post-ViE Phase (N=14)
Hypotension (Vascular disorders) | 11 (27) | 12 (110) | 9 (28)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (11) | 11 (26) | 2 (3)
Fluid Overload (Metabolism and nutrition disorders) | 4 (5) | 11 (28) | 3 (4)
Dizziness (Nervous system disorders) | 5 (6) | 7 (13) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less